CLINICAL TRIAL: NCT07240779
Title: Evaluating the Use of Advanced Sperm Selection Methods on ICSI Procedure Outcomes by Physiological Intracytoplasmic Sperm Injection (PICSI) Verses ZyMot Device
Brief Title: Advanced Sperm Selection in ICSI: A Comparative Study of PICSI and ZyMot
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunrise Fertility Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PICSI-ZYMOT methods
Record Dates: First submitted 2025-09-25; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Infertile Patient Undergoing ICSI Procedure
Keywords: ICSI; PICSI; ZYMOT

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ICSI group (No Intervention): Sperm selection performed using traditional methods
- : PICSI Group (Active Comparator): * Sperm selection performed using the Physiological Intracytoplasmic Sperm Injection (PICSI) method.
  * Hyaluronic acid-based selection to choose mature, DNA-intact sperm.
  * Followed by standard ICSI procedure.
  Interventions: Device: picsi dish
- ZyMot Group (Active Comparator): * Sperm selection performed using the ZyMot microfluidic device.
  * Mimics natural sperm migration to isolate motile, morphologically normal sperm.
  * Followed by standard ICSI procedure
  Interventions: Device: picsi dish

INTERVENTIONS:
Device: picsi dish — theses techniques to selection mature and lowest DNA fragmentation sperm for injection in oocyte
  Other Names: zymot device
  Arms: : PICSI Group; ZyMot Group

SUMMARY:
our study explores the effectiveness of two advanced sperm selection techniques-PICSI and the ZyMot microfluidic device-in improving outcomes of Intracytoplasmic Sperm Injection (ICSI). It aims to compare their impact on fertilization rates, embryo quality, and clinical pregnancy success, helping determine which method offers superior results in assisted reproductive technology.

ELIGIBILITY:
Inclusion criteria:-

* Age for women is between 20-39 years old.
* Body mass index (BMI) between 19 kg/m and 35 kg/m
* Normal Prolactin level.
* No other endocrinological abnormality including thyroid disorder or diabetes.
* With antimullerian hormone (AMH) at least 1.5 ng/ml, ), with normal progesterone level.
* Primary or secondary infertility at least of 2 years duration.
* No evidence of endometriosis.
* No other medical or surgical disease.
* The day of embryo freezing is the fifth day (day 5), and all patients who undergo the process of transferring frozen embryos.
* The endometrium thickness is between 8-14 mm on day of transfer.
* Inclusion criteria of male partner were; presence of ejaculate motile spermatozoa with total sperm number 1 million/ml at least and sperm motility 5% or more and all patient with high DNA fragmentation index above 35%.

Exclusion criteria׃-

* Women were older than 40 years of age or younger than 18 years old.
* Women laparoscopically diagnosed to have endometriosis within the last 1 year.
* Male infertility factor with immotile sperm.

Ages: 20 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Primary outcome measure | 6-9 weeks after embryo transfer.
  1• clinical pregnancy rate:- defined as the presence of a fetal heartbeat or gestational sac.
  • Unit of Measure: Percentage (%)

SECONDARY OUTCOMES:
secondary outcome measure | 1-After 6 weeks of gestation.
  1- Miscarriage rate: Defined as pregnancy loss following confirmation of clinical pregnancy. Unit of Measure: Percentage (%)

CONTACTS AND LOCATIONS:
Overall Officials: Ayat samir kamel, Principal Investigator — Sunrise Fertility Center; Rafaat Gabre, phd, Study Director — faculity of science, Cairo university; Omaima Idris, phd, Study Director — faculity of medicien, cairo university; Abeer mohsen, Study Chair — faculity of science, cairo University; Ahmed Said, Study Chair — Faculty of Science, Al-Azhar University, Assiut